CSMC Date Effective: 10/4/2022



TITLE: PHASE IB/II TRIAL OF ANTI-PD-1 IMMUNOTHERAPY AND STEREOTACTIC RADIATION IN PATIENTS WITH RECURRENT GLIOBLASTOMA

STUDY SUPPORT PROVIDED BY: CEDARS-SINAI MEDICAL CENTER; NATIONAL INSTITUTES OF HEALTH; MERCK & CO., INC.

PRINCIPAL INVESTIGATOR: CHIRAG PATIL, MD

STUDY CONTACT PHONE NUMBER AT CSMC: 310-248-6693

**AFTER HOURS CONTACT (24 HOURS): 310-423-7900** 

This research study is sponsored by Cedars-Sinai Medical Center and National Institutes of Health, with study drug support provided by Merck & Co., Inc. Merck & Co., Inc. only reimburses Cedars-Sinai Medical Center for the costs associated with running the study; Merck & Co., Inc. is not providing additional compensation to Cedars Sinai Medical Center or the Principal Investigator for their participation in the study.

#### 1. WHAT IS THE PURPOSE OF THIS RESEARCH STUDY?

We are doing this study to see if pembrolizumab (study drug) combined with standard of care stereotactic radiation therapy and surgery is safe and effective in patients with recurrent glioblastoma. We will give pembrolizumab and radiation to research participants and watch carefully for any side effects. We want to know if giving pembrolizumab is safe, tolerable, and feasible, and whether it improves overall survival, increases the length of time during and after treatment that your cancer does not get worse, and to evaluate how well the body responds to a treatment.

You are being asked to take part in this research study because you have glioblastoma with recurrence or progression and are planning to undergo standard of care stereotactic radiation therapy and surgical resection.

The study will enroll up to 30 people in total.

This research study is designed to test the investigational use of pembrolizumab. This drug is approved by the U.S. Food and Drug Administration (FDA) for some skin, lung, head and neck, hematological (lymphoma), urological (kidney and bladder), gastrointestinal (liver, stomach, esophagus, and colon), breast gynecological cancers (lining of the uterus and cervical) and it is also used for cancers whose tumor cells have special features. However, it is not approved by the FDA for glioblastoma.

CSMC Date Effective: 10/4/2022

# 2. WHAT WILL HAPPEN DURING THE STUDY?

This section provides a general overview of what will happen during your participation in this study. Information included below should be considered along with the flowchart of procedures attached as an Appendix.

The flowchart shows a timeline for research-related or standard of care procedures that are involved in your participation in this study. **Research-related procedures** are those performed solely for the research. They would not be performed if you did not take part in the study. **Standard of care** (**routine**) procedures would be performed both as part of this study and if you do not participate in this study.

A table describing common medical procedures done solely for the purposes of monitoring and assessing your condition during this study is attached as an Appendix to the end of this consent form. Standard of care procedures that will be repeated or done at greater frequency are listed in the flow chart Appendix.

#### Overview of study:

If you choose to participate in this study, you will receive one dose of the study drug intravenously (through the vein) before your planned radiation therapy and surgery. After surgery, you will receive study drug infusions every 6 weeks until disease progression, intolerable side effects, withdrawal of consent, or up to 2 years or 18 cycles of study drug, whichever comes first. In addition, research blood will be collected at five time points during the study, and fresh research tumor specimens will be collected at your standard of care surgical resection. Additional tumor tissue will be obtained from the fresh tumor specimen later to be used for research purposes.

These research blood and tumor samples will be collected in order to evaluate biomarkers (made of DNA, RNA, proteins, cells or components of cells). A biomarker is a biological molecule found in blood, other body fluids, or tissues that may be a sign of a condition or disease. Biomarkers also involve studies of your genes (DNA) and studies will be done to see whether differences in genes are associated with activity of the study drug or if genes change over time. These samples will not be used to make decisions about your eligibility, treatment assignment, or other clinical management. They will only be used for research to learn more about the disease and how it responds to treatment.

This study requires you to stop certain treatments for 1-4 weeks so they may be flushed from your body in order to prevent conflicts with the study drug. For this study, you are required to stop taking cancer therapies (except temozolomide) including any investigational (not FDA approved) drugs for 4 weeks and stop receiving certain radiation therapy for 1 week. Consult with the researchers before taking any non-study medications including over-the-counter drugs or vitamins. Possible risks from the washout are discussed in the section "What are the Possible Risks or Discomforts?"

In order to properly follow the study's protocol (research plan), all participants will receive treatments and procedures that have been pre-determined by the protocol. In effect, the protocol describes which medications or procedures you will receive, rather than those decisions being made

CSMC Date Effective: 10/4/2022

by your personal doctor or based on your preference. There may be options available outside of this study that you will not be able to receive while participating in this study. We do not believe you should be at any increased risk due to this limitation.

Treatments for your disease can cause side effects. If you experience side effects, you will receive medications to help deal with these side effects and may need additional procedures to evaluate the side effects. The drugs or procedures you may receive are given as part of routine care for side effects.

#### How long will you be in the study?

We think you will be in this study for about 6 months on average. The total time includes about 1 month of screening, about 1 month of treatment through surgery (including 1 day of treatment with the study drug, 3 days of radiation therapy, and 1 day of surgery), and approximately 4 months of treatment (on average) following surgery. After that, we would like you to keep in touch with you every 2 months, via medical record review, telephone contact, or in-clinic contact, to see how you are doing.

# 3. WHAT ARE THE POSSIBLE RISKS?

Risks of common medical procedures performed solely for research purposes are described in a table attached to the end of this consent form as an Appendix. Side effects and risks of standard of care procedures are not described in this consent form.

This section describes the possible risks and/or discomforts we anticipate you could experience that are related to the study procedures.

#### **Unknown Risks**

There may be other side effects or risks that we cannot predict. Many side effects may go away shortly after the study medication or procedure is stopped. However, in some cases they can be serious, long-lasting, permanent, and/or fatal.

#### Risks of Pembrolizumab

Pembrolizumab works by helping your immune system to fight your cancer. However, pembrolizumab can also cause your immune system to attack normal organs and tissues in your body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e. causing hospitalization or be life-threatening), may result in death, and/or may occur after you stop taking pembrolizumab. These side effects can affect more than one of your normal organs and tissues at the same time.

#### **VERY COMMON**

Out of 100 people who receive pembrolizumab, 20 or more people may have the following:

- Itching of the skin
- Loose or watery stools
- Cough
- Fatigue
- Muscle/joint pain
- Decreased appetite
- Nausea

CSMC Date Effective: 10/4/2022

Rash

• Fever

#### **COMMON**

# Out of 100 people who receive pembrolizumab, at least 5 but less than 20 people may have the following:

- Back pain
- Pain in your belly
- Loss of skin color
- Not enough thyroid hormone so you may feel tired, gain weight, feel cold, or have infrequent or hard stools (hypothyroidism)
- Low levels of salt in the blood that may cause you to feel tired, feel confused, have a headache, have muscle cramps, and/or feel sick to your stomach (hyponatremia)
- Shortness of breath
- Constipation
- Headache
- Vomiting
- Anemia (low levels of red blood cells)
- Swelling of the arms and legs

#### **UNCOMMON**

# Out of 100 people who receive pembrolizumab, at least 1 but less than 5 people may have the following:

- Inflammation of the lungs, so you may feel short of breath and cough (pneumonitis)
- Too much thyroid hormone, so you may feel anxious, feel angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools (hyperthyroidism)
- Infusion reaction, where you may feel dizzy or faint, feel flushed, get a rash, have a fever, feel short of breath, experience a decrease in your blood pressure at the time of receiving your infusion (IV) or just after, or have pain at the site of infusion
- Inflammation of the bowels/gut, which may cause severe pain in your belly with loose or watery stools, and black, tarry, sticky stools or stools with blood or mucus (colitis)
- Inflammation of the skin so you may have peeling of the skin, itchiness, and/or skin redness. The skin inflammation (i.e., peeling, itching and redness) could also be widespread throughout your body. More severe skin reactions may involve the inside of your mouth, the surface of your eye and genital areas, and/or may cause the top layer of your skin to peel from all over your body which can cause severe infection (Severe skin reactions, including Stevens-Johnson syndrome/or toxic epidermal necrolysis)

#### RARE

# Out of 100 people who receive pembrolizumab, less than 1 person may have the following:

- Inflammation of the nerves that may cause pain, weakness, or tingling in your hands and feet, and may spread to your legs, arms, and upper body, leading to severe muscle weakness and possible temporary paralysis (Guillain-Barré syndrome)
- Inflammation of the muscles, so you may feel weak or have pain in your muscles (myositis)

CSMC Date Effective: 10/4/2022

• Inflammation of the pancreas (a gland in your abdomen that controls sugar levels), so you may have severe pain in the top part of your belly that may move to your back, feel sick to your stomach, and have vomiting that gets worse when you eat (pancreatitis)

- Inflammation of the eye, so you may have eye redness, blurred vision, sensitivity to light, eye pain, see floaters, or have headaches (uveitis)
- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, a pain in the right side of your belly, yellow eyes and skin, and dark urine (hepatitis)
- Inflammation of the pituitary gland (a gland in the head), which may cause you to feel sick to your stomach or have headaches, changes in your behavior, double vision, few to no menstrual cycles, weakness, vomiting and dizziness, or fainting (hypophysitis)
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone, which could cause tiredness, weight loss, muscle weakness, feeling faint, having joint, muscle, and belly aches, nausea, vomiting, loose or watery stools, fever, salt craving, and sometimes darkening of the skin like a suntan (adrenal insufficiency)
- Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination, and weight loss. You are likely to need regular insulin shots
- Inflammation of the kidney, so you may pass less urine or have cloudy or bloody urine, swelling, and low back pain (nephritis)
- Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath, and swelling of the legs. You may experience a fast or irregular heartbeat that may cause dizziness or fainting (myocarditis)
- Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy (thyroiditis)
- A condition that may make you feel weak and tired and may cause drooping of the eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your arms and legs, or difficulty breathing (myasthenic syndrome/myasthenia gravis including exacerbation)
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin, or lungs (sarcoidosis)
- Inflammation of the brain with confusion and fever. This may also include: disorientation, memory problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of movement in some parts of your body, and loss of consciousness (encephalitis)
- Inflammation of the spinal cord with pain, numbness, tingling, or weakness in the arms or legs, bladder or bowel problems including needing to urinate more frequently, urinary incontinence, difficulty urinating, and constipation (myelitis)
- Inflammation of the blood vessels (vasculitis). Symptoms will depend on the particular blood vessels that are involved in the inflammatory process, for example; if it is your skin, you may get a rash. If your nerves are not getting enough blood, you could have numbness and weakness. You may also experience fever, weight loss, and fatigue.
- Low levels of parathyroid hormone (a hormone made by 4 tiny glands in your neck) which may result in low blood calcium and cause muscle cramps or spasms; fatigue or weakness; numbness, tingling or burning in your fingertips, toes or lips (hypoparathyroidism)

CSMC Date Effective: 10/4/2022

Additionally, since pembrolizumab was approved in September 2014, the following side effects have been reported by people receiving pembrolizumab. These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of these side effects:

- Inflammation of the joints which may include joint pain, stiffness and/or swelling (arthritis)
- Severe responses of the immune system that cause the body to attack its own blood cells, spleen, liver, lymph nodes, skin and brain. This may include fever, rash, inflammation of the liver, yellowing of the skin, an enlarged liver and spleen, low blood counts, and enlarged lymph nodes. The nervous system may also be affected and cause confusion, seizures, and even coma (hemophagocytic lymphohistiocytosis)
- Changes in eyesight, eye pain, whitish patches on the skin and hearing loss (Vogt-Koyanagi-Harada syndrome)
- Inflammation and scarring of the bile ducts (tubes that carry digestive fluid that is made in the liver). This can cause symptoms similar to those seen with inflammation of the liver (hepatitis) such as pain in right side of your belly, yellow eyes and skin, feeling tired, and itching (sclerosing cholangitis).

If you have had an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), you may experience graft versus host disease (GvHD), which may include diarrhea, skin rashes, and liver damage, after receiving pembrolizumab. Sometimes this condition can lead to death.

If you have had a solid organ transplant (for example, if you have received a kidney or heart transplant), you may experience rejection of the transplanted organ. Your doctor will monitor you and should tell you what signs and symptoms you should report depending on the type of organ transplant that you have had.

#### Reproductive and Lactation Risks

Taking part in this research study can affect an unborn baby. Therefore, you should not become pregnant or father a baby while on this study. If you or your partner is capable of becoming pregnant you will need to use birth control throughout the study and for at least four (4) months after the last dose of study drug. Check with the researcher about approved birth control methods to use while participating in this study.

Women should not breastfeed a baby while on this study.

#### *Unknown Risks to the Developing Embryo or Fetus (an unborn baby)*

If you are pregnant, or become pregnant during participation in this research, the study drug, procedures, or radiation might involve risks to an embryo or fetus, which are currently unknown. It is important that you contact the researcher immediately if you believe you might be pregnant.

#### Collection of Pregnancy Outcomes

If you become pregnant during the study, we will collect information on the outcome of your pregnancy including spontaneous or voluntary termination, details of the birth, and the presence or absence of any birth defects, abnormalities, or complications, and the health status of your child. By signing this consent, you are agreeing to have this information about you and your child collected from your medical records in the rare case that you become pregnant during your participation in this research study, however, you are always free to withdraw your consent to participate in any research procedure.

CSMC Date Effective: 10/4/2022

#### Risks of Discontinuation of Current Medication

In order to participate in this research study, you must stop taking live vaccines and any medications you are currently taking for your cancer. This may result in a worsening of your condition. Your physician will continuously monitor your condition to determine whether it is safe for you to continue in this study.

#### Follow-up Visit for Discontinuing Participants

While you are free to discontinue your participation at any time, we encourage you to complete a Final Study Visit. During this visit, we will conduct tests to collect safety data, and discuss any information that may be important to share with your treating physician.

#### 4. ARE THERE BENEFITS IN TAKING PART IN THE STUDY?

If you agree to take part in this research study, there may or may not be direct medical benefit to you. The possible benefit of taking part in the research study is that it may help you live longer. However, no benefit is guaranteed. It is possible that your condition may remain unchanged or even get worse.

We hope the information learned from this research study will benefit other individuals with glioblastoma in the future by helping us to learn whether taking pembrolizumab prior to and after radiation and surgery is safe and whether it improves survival outcomes and the body's immune response.

### 5. WILL I BE INFORMED OF RESEARCH RESULTS?

Some of the research tests done in this study follow standard clinical procedures and are performed in certified clinical labs. These test results may be shared with you and may be placed in your Cedars-Sinai medical record. Other research tests done in this study are for research purposes only and are performed in a research only lab where the results are not intended for clinical use. These research-only results will not be shared with you or included in your Cedars-Sinai medical record.

#### **Unanticipated Incidental Findings**

If, unexpectedly, we find that results of your research procedures could suggest important medical information and we determine there is something you or your doctors can do in response to this finding, we will contact you using the last contact information provided by you. If necessary, we may recommend additional clinical testing to confirm the research finding. The cost of any additional testing and any related treatment will be your responsibility.

# 6. WHY WOULD MY PARTICIPATION BE STOPPED?

Your participation in this study may be stopped at any time by the researcher or the sponsor without your consent for any reason, including:

- The study is stopped or suspended;
- Funding for the study is reduced, stopped or withdrawn;
- If it is in your best interest;
- You do not consent to continue in the study after being told of changes in the research that may affect you;

CSMC Date Effective: 10/4/2022

• You do not follow the study procedures.

You may choose (or you may be required) to withdraw from certain parts of the study, but invited to continue with other parts. For example, you might stop taking a study drug, but continue with follow-up visits or allow us to continue to collect data from your medical records. Separate written consent will be requested if your continued participation will involve procedures not described in this consent form.

# 7. ARE THERE ANY OTHER OPTIONS?

Your participation is voluntary, so you have the right to decline to participate or to withdraw from this research study at any time without any penalty or loss of benefits to which you would be entitled outside of the study. Choosing not to participate will not affect the care you receive at Cedars-Sinai Health System.

If you decide not to take part in this study, you have other choices. For example:

- you may choose to be treated following the usual clinical approach, such as radiation therapy and surgery without the addition of the study drug, pembrolizumab
- you may choose to take part in a different study at CSMC or elsewhere, if one is available
- you could decide not to be treated.
- you may choose to pursue supportive or palliative care for your condition. Such care is focused on reducing suffering and improving the quality of life of individuals with chronic or life-threatening illnesses. The primary intent of palliative care is not to cure a disease or to prolong life. Palliative therapy is focused primarily on managing symptoms.

The researcher will discuss these options and their risks and benefits with you.

# 8. WILL MY INFORMATION BE KEPT CONFIDENTIAL?

We will do our best to make sure that the personal information collected as part of this study is kept private. However, we cannot guarantee total privacy. A copy of your research consent and authorization forms may be filed in your electronic medical record at CSMC. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other identifiable personal information will not be used. Organizations that may look at and/or copy your medical records for research oversight, quality assurance, and data analysis include: accrediting agencies, government and regulatory groups (such as Food and Drug Administration (FDA), Office for Human Research Protections (OHRP), etc.), safety monitors, companies that sponsor the study, and authorized representatives of the sponsor.

Attached to this consent form is an "Authorization Form" that outlines with whom your information may be shared for the purposes of this research and under what circumstances.

We might share your information and/or research samples collected in this study with other researchers at Cedars-Sinai, other academic institutions, or third party commercial entities for future research without additional informed consent from you. Information that identifies you will be removed and will not be shared with other researchers or anyone outside of Cedars-Sinai.

CSMC Date Effective: 10/4/2022

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

# Protections From Forced Disclosures (Subpoenas) - Certificates of Confidentiality

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence, unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate does not stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases and threats to harm yourself or others. The Certificate cannot be used to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate does not stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also does not prevent your information from being used for other research, if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

#### 9. WHAT IF I BECOME ILL OR INJURED BECAUSE OF TAKING PART IN THIS STUDY?

Contact your study doctor at once if you feel that you are ill or have been injured because of taking part in this study. If it is a medical emergency, call 911 or go to an emergency room. Promptly notify your study doctor of your situation at the phone number listed on page 1 of this consent form.

# Who pays for my research related illness or injury?

Cedars-Sinai has no plans to pay for costs associated with the treatment of research-related injury or illness. We will make every effort to seek reimbursement from your health plan. However, you will be responsible for any deductibles and co-payments required under your health plan and for any claims ultimately denied by your health plan. Financial assistance may be available under Cedars-Sinai's Charity Care Policy and Procedure. If you feel that you have had a research-related injury and need financial assistance, please contact the IRB Office at 310-423-3783. You do not waive any of your legal rights by signing this form.

#### 10. FINANCIAL CONSIDERATIONS

#### Costs of Participation

Please review the attached Appendix flowchart for a listing of items, drugs and services that will be billed to you and/or your insurance and those that will be covered by the study sponsor.

CSMC Date Effective: 10/4/2022

Only items, drugs and services that are reasonable and necessary for your medical care throughout the study will be billed to your insurance. You remain responsible for all deductibles, co-pays, and balances under your health benefit plan. If your insurance company does not pay, you will be billed for those charges. You should check with your health benefit plan if you have questions or concerns about your insurance coverage.

#### Compensation for Participating

You will not be paid for taking part in this research study.

#### Financial Interest in the Research

The PI and institution have no potential financial conflict of interest with respect to this study.

# 11. WHAT IF I HAVE QUESTIONS OR PROBLEMS?

Please contact the investigator listed on the first page of this form for questions or concerns about the research.

If you have questions, problems, or concerns that you want to discuss with someone who is not associated with this study, or want to offer suggestions or feedback, please contact:

Cedars-Sinai Human Research Protection Program (HRPP) Phone: (310) 423-3783 Email: ResearchConcerns@cshs.org

The Cedars-Sinai HRPP has been established to protect the rights and welfare of research participants. You may also contact the Cedars-Sinai HRPP if you want to offer input or obtain information regarding the study.

#### 12. CONSENT PROVISIONS

If you sign this form below, it means that:

- (1) You have taken the time to carefully read and understand the information presented in this informed consent form; you should discuss it with others, and if appropriate seek a second opinion to make an informed decision;
- (2) The information concerning the research study and its involved procedures has been fully explained to you and your questions have been answered to your satisfaction;
- (3) You have received and understand all of the information you desire regarding your participation in the research study;
- (4) You have considered the potential risks, any anticipated benefits and alternatives (and their relative risks and benefits) of participation;
- (5) You are voluntarily agreeing to participate in this research study;
- (6) You understand that by consenting to participate in the research, you are not giving up any of your legal rights;
- (7) You understand that you have the right to be informed of significant new findings related to this research study which may affect your willingness to continue participating in this study; and
- (8) You have been provided with a copy of the "Experimental Subject's Bill of Rights", if applicable to this research study, and have been provided with an opportunity to ask questions regarding the Bill of Rights.

CSMC IRB No: STUDY00001234 / MOD00006302 CSMC Date Effective: 10/4/2022

We will give you a copy of this signed and dated consent form and the Experimental Subject's Bill of Rights.

CSMC IRB No: STUDY00001234 / MOD00006302 CSMC Date Effective: 10/4/2022

# SIGNATURE PAGE

# **Consent Form for Research and Authorization for Use and Disclosure of Identifiable Health Information (Research)**

| SIGNATURE BY THE PARTICIPANT: I hereby agree to participate in the research study described to me during the informed consent process and described in this informed consent form. You will be given a signed copy of this form. | | |
|---|---|---|
| Name of Participant (Print) | Signature | Date Signed |
| Authorization for Use and Disc (Research): I hereby agree that and/or disclosed in accordance will dentifiable Health Information (Association) | ny identifiable health inf<br>yith this "Authorization f | formation may be used for Use and Disclosure of |
| Name of Participant (Print) SIGNATURE BY THE INVESTIGA described in this form have been discus further attest that all questions asked b | ssed fully in non-technical ter | rms with the participant. I |
| Name of Investigator (Print) | Signature | Date Signed |
| SIGNATURE BY THE INTERPRET (Signature of an interpreter is only requith the assistance of an interpreter and person who is conversant in both English such as the interpreter (the certified hoperson. The witness signs the consent) | TER/WITNESS uired when a non-English sp id an IRB-approved 'short fo ish and the language of the N ospital interpreter), study staj | eaking subject is consented<br>rm.' The witness may be any<br>Ion-English speaking subject,<br>ff, a family member, or other |
| Name of Witness (Print) | Signature | Date Signed |

CSMC Date Effective: 10/4/2022



# APPENDIX: EXPERIMENTAL SUBJECT'S BILL OF RIGHTS

In accordance with California Health and Safety Code 24172, any person who is required to consent to participate as a subject in a research study involving a medical experiment or who is requested to consent on behalf of another has the right to:

- 1. Be informed of the nature and purpose of the experiment.
- 2. Be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized.
- 3. Be given a description of any attendant discomforts and risks to the subject reasonably to be expected from the experiment.
- 4. Be given an explanation of any benefits to the subject reasonably to be expected from the experiment, if applicable.
- 5. Be given a disclosure of any appropriate alternative procedures, drugs or devices that might be advantageous to the subject, and their relative risks and benefits.
- 6. Be informed of the avenues of medical treatment, if any, available to the subject after the experiment if complications should arise.
- 7. Be given an opportunity to ask any questions concerning the experiment or the procedure involved.
- 8. Be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation in the medical experiment without prejudice.
- 9. Be given a copy of any signed and dated written consent form used in relation to the experiment.
- 10. Be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion, or undue influence on the subject's decision.

CSMC Date Effective: 10/4/2022



# <u>AUTHORIZATION FOR USE AND DISCLOSURE OF</u> IDENTIFIABLE HEALTH INFORMATION FOR RESEARCH

# USE AND DISCLOSURE OF HEALTH INFORMATION

If you agree to this Authorization, you give permission to the Sponsor, Principal Investigator, other investigators and their research team described in the Consent Form for Research ("Research Team") to use or disclose your identifiable health information ("private information") for the research study titled "PHASE IB/II TRIAL OF ANTI-PD-1 IMMUNOTHERAPY AND STEREOTACTIC RADIATION IN PATIENTS WITH RECURRENT GLIOBLASTOMA" which is described in the Consent Form for Research ("Consent Form") to which this Authorization is attached. In particular, you authorize the research team acting under the direction of the Principal Investigator to review your medical records and collect your private information from the following sources:

| ■ Laboratory tests | ☑ Doctor/clinic records |
|---|---|
| ☐ Pathology reports | ☑ Hospital/medical records |
| ☐ Imaging reports (e.g., x-rays or scans) | ☐ Mental health records |
| ☑ Photographs or videos of your image | ☐ Billing records |
| ☑ Other tests or other types of medical inf | formation: electrocardiogram results |

# • WHO WILL HAVE ACCESS TO YOUR PRIVATE INFORMATION?

Your private information will be used by and/or shared with the Research Team.

In addition to the research team, if applicable, the following parties may receive your private information and inspect your records:

- The reviewing Institutional Review Boards and Cedars-Sinai offices with authority to oversee research compliance.
- U.S. government agencies, such as the Food and Drug Administration and the Department of Health and Human Services.
- Researchers at other organizations who are participating in this research study.
- The Study Sponsor, its business partners, and Cedars-Sinai's business partners for matters related to research study oversight, data analysis and use of research results in product development, and payment or reimbursement.

CSMC Date Effective: 10/4/2022

• Representatives from regulatory agencies in other countries may join in the review of your research records, including research-related medical reports and information, with the Sponsor and/or the FDA.

Cedars-Sinai is required by law to protect your private information. However, the recipients described above may re-disclose (or share) your information with other parties unless such sharing is prohibited by law.

# • WHEN WILL MY AUTHORIZATION EXPIRE?

By signing this document, you authorize the use and sharing of your private information until the end of the research study and any related optional sub-study you choose to participate in.

# REVOKING AUTHORIZATION

You may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, the research team may still use or disclose private information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. To revoke this Authorization, you must write to the Principal Investigator of the research study by writing to the Office of Research Compliance and Quality Improvement, 6500 Wilshire Blvd, Suite 1800, Los Angeles, Calif. 90048 and/or emailing to ResearchConcerns@cshs.org.

# • NOTICE OF RIGHTS AND OTHER INFORMATION

You do not have to agree to this Authorization, but if you do not agree, you may not participate in the research study. The Research Team may not condition (withhold or refuse) treating you on whether you agree to this Authorization.

If you agree to this Authorization, please sign on the appropriate signature line on the Signature Page. You will receive a copy of this Authorization.

CSMC Date Effective: 10/4/2022

# APPENDIX: Detailed Description of Common Medical Procedures Performed for Research Purposes and Associated Risks

The procedures listed below are often performed as part of routine care for a person with your condition. They are being repeated, or performed more frequently as part of this research. However, the risks associated with each procedure should be comparable to what you would experience even if you were undergoing the procedure outside this research study.

| Study Procedure | Related Risks |
|---|---|
| <b>Blood draw:</b> A needle is placed in the vein in your arm to draw blood | Blood drawing may cause some pain and has a small risk of bleeding, bruising, or infection at the puncture site. There is also a small risk of fainting. |
| Electrocardiogram (ECG): abbreviated as EKG or ECG – is a test that measures the electrical activity of the heartbeat using electrodes (disposable adhesive discs placed on the skin). | There's no pain or risk associated with having an electrocardiogram. When the disposable adhesive discs are removed from your skin, there may be some minor skin discomfort or irritation. You may experience temporary discomfort (pulling on the skin/skin hair) during removal of the patches. This hair may be shaved for patch placement. |
| Infusion Procedure: Infusion is the administration of drugs directly into your bloodstream using intravenous (IV) lines. The risks associated with IV lines are described separately below. | Occasionally, people have allergic reactions (including life-threatening reactions) when taking any medication. Symptoms of any allergic reaction can include a rash, hives, itching, and/or difficulty breathing, closing of the throat, swelling of the lips, tongue or face, and rarely death. If you experience any difficulty breathing, closing of the throat, swelling of the lips, tongue or face, or hives, you should stop taking your study drug and immediately seek emergency medical attention. |
| | In general, allergic reactions to medicines are more likely to occur in people who have allergies to other drugs, foods, or things in the environment, such as dust or grass. If you have allergies to other medicines, foods, or other things in the environment, or if you have asthma, you should let your researcher know. |
| Intravenous (IV) lines: You will receive the study drug or other medications or contrast agent through an intravenous (IV) line. An IV line is a small tube that is attached to a catheter and inserted by needle into a vein usually in your hand or arm. Qualified medical professionals will place IV lines for use in this study. | IV lines are usually safe and well tolerated and complications are rare, but can include phlebitis (swelling of the vein) and infection. The IV may come out accidentally or blood may leak around the line. If the IV is not in the vein, medication or fluid can enter the surrounding soft tissues, and can be associated with swelling, discomfort, bruising and irritation. Rarely, a clot can develop in the IV line itself. If this happens, the staff may |

CSMC IRB No: STUDY00001234 / MOD00006302 CSMC Date Effective: 10/4/2022

| | remove the old IV line and start a new IV line. There is also a small risk of feeling lightheaded and fainting. |
|---|---|
| Magnetic Resonance Imaging (MRI): A | You may feel slightly anxious inside the scanner |
| MRI is a test that uses a magnetic field and | due to a fear of small enclosed spaces |
| pulses of radio wave energy to make pictures | (claustrophobia). Also, at times, you may hear |
| of organs and structures inside the body. | very loud noises as the MRI machine is taking |
| During the procedure you will lie down in a | pictures of your body. You may be given |
| large donut-like looking magnet and we will | headphones and may request ear plugs if you feel |
| ask you to lie still on a table for the duration | the noise is too loud. At any time, you may ask |
| of the procedure (about 2 hours). You will be | the technician to stop the exam if you are unable |
| able to communicate with researchers all the | to complete the exam. |
| time and you will have a panic button to use | |
| if you want to stop the procedure at any time. | |
| Physical Exam: Includes height, weight, | There are no physical risks associated with these |
| vital signs (heart rate and blood pressure) | procedures. |
| Concomitant Medications: You will be | There are no physical risks associated with these |
| asked about your previous and current | procedures. |
| medications that you take. | |
| Medical History Review: You will be asked | There are no physical risks associated with this |
| about your medical and surgical history with | procedure. |
| attention to [Insert as appropriate: smoking | |
| and alcohol habits, menopausal history | |
| (females only) and your physical activity] | |
| <b>Pregnancy Test:</b> If you are a woman who is | If your test is positive, you will be told and at that |
| able to become pregnant, [blood/urine] | point you should discuss options available with |
| samples will also be used to do a pregnancy | your primary physician. |
| test | |
| <b>Demographic Information:</b> You will be | There are no physical risks associated with these |
| asked about your age, gender, race, ethnicity | procedures. |